CLINICAL TRIAL: NCT01624571
Title: A Double-blind, Multi-center, Randomized, Placebo-controlled, Parallel, Phase II Clinical Trial to Assess the Effect on Recovery of GI Motility and Safety and to Determine the Optimal Dose of LD02GIFRO in Patients Undergoing Colon Resection
Brief Title: Study to Assess the Effect on Recovery of GI Motility and Safety and to Determine the Optimal Dose of LD02GIFRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LG-GRCL001
Record Dates: First submitted 2012-06-07; First posted 2012-06-20 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2012-10

CONDITIONS: Colon Resection; _large Interstinal Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): 300mg/day
  Interventions: Drug: LD02GIFRO
- Group 2 (Experimental): 600mg/day
  Interventions: Drug: LD02GIFRO
- Group 3 (Experimental): 900mg/day
  Interventions: Drug: LD02GIFRO
- Placebo (Placebo Comparator): Control Group
  Interventions: Drug: LD02GIFRO

INTERVENTIONS:
Drug: LD02GIFRO — comparison of different dosages of drug

SUMMARY:
This clinical trial is conducted to determine the optimal dose of LD02GIFRO in improvement of gastrointestinal motility between each dose group by comparing the effectiveness and safety in patients undergoing colon resection.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 20 years
* Subject is scheduled for a partial colon resection with primary anastomosis via laparotomy
* Subject is scheduled to receive primary postoperative pain management with intravenous patient-controlled analgesia (PCA) opioids

Exclusion Criteria:

* Subject is scheduled for a total colectomy, colostomy, ileostomy
* Subject has complete bowel obstruction
* Subject is scheduled for laparoscopic surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Improvement of gastrointestinal motility | in hospitalization (Maximized 14 days)
  Evaluation gastrointestinal function to the time of improvement gastrointestinal motility

CONTACTS AND LOCATIONS:
Locations (1):
- Asan medical center, Seoul, South Korea